CLINICAL TRIAL: NCT02347176
Title: A Phase 2b, Randomized, Double-blinded, Placebo-controlled, Dose-ranging Study to Evaluate the Efficacy and Safety of Tralokinumab in Adult Subjects With Moderate-to-Severe Atopic Dermatitis
Brief Title: Phase 2 Study to Evaluate the Efficacy and Safety of Tralokinumab in Adults With Atopic Dermatitis
Acronym: D2213C00001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2213C00001
Record Dates: First submitted 2015-01-05; First posted 2015-01-27 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo matched to Tralokinumab will be administered subcutaneously to participants once every 2 Weeks (Q2W) for 12 weeks.
  Interventions: Other: Placebo
- Tralokinumab Dose 1 (Experimental): Tralokinumab Dose 1 will be administered subcutaneously once every 2 Weeks (Q2W) for 12 weeks.
  Interventions: Biological: Tralokinumab Dose 1
- Tralokinumab Dose 2 (Experimental): Tralokinumab Dose 2 will be administered subcutaneously once every 2 Weeks (Q2W) for 12 weeks.
  Interventions: Biological: Tralokinumab Dose 2
- Tralokinumab Dose 3 (Experimental): Tralokinumab Dose 3 will be administered subcutaneously once every 2 Weeks (Q2W) for 12 weeks.
  Interventions: Biological: Tralokinumab Dose 3

INTERVENTIONS:
Other: Placebo — Subcutaneous injection with placebo
  Arms: Placebo
Biological: Tralokinumab Dose 1 — Subcutaneous injection with tralokinumab
  Arms: Tralokinumab Dose 1
Biological: Tralokinumab Dose 2 — Subcutaneous injection with tralokinumab
  Arms: Tralokinumab Dose 2
Biological: Tralokinumab Dose 3 — Subcutaneous injection with tralokinumab
  Arms: Tralokinumab Dose 3

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of tralokinumab in adults with atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of atopic dermatitis for greater than (>) 1 year
* Atopic dermatitis involvement of greater than or equal to (>=) 10 percent (%) body surface area
* EASI score of >= 12
* SCORAD of >= 25
* IGA score of >= 3
* Effective birth control in line with protocol details

Exclusion Criteria:

* History of anaphylaxis following any biologic therapy
* Hepatitis B, C or human immunodeficiency virus
* Pregnant or breastfeeding
* History of cancer
* Previous receipt of tralokinumab

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2015-01-23 (Actual); Primary Completion 2015-11-27 (Actual); Study Completion 2016-02-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (52):
- United States (22):
  - Research Site, Phoenix, Arizona
  - Research Site, Rogers, Arkansas
  - Research Site, Fremont, California
  - Research Site, Fullerton, California
  - Research Site, Los Angeles, California
  - Research Site, Oceanside, California
  - Research Site, Rancho Santa Margarita, California
  - Research Site, Santa Monica, California
  - Research Site, Clearwater, Florida
  - Research Site, Miami, Florida
  - Research Site, Worcester, Massachusetts
  - Research Site, Warren, Michigan
  - Research Site, Berlin, New Jersey
  - Research Site, Verona, New Jersey
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Portland, Oregon
  - Research Site, Charleston, South Carolina
  - Research Site, Houston, Texas
  - Research Site, Pflugerville, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Norfolk, Virginia
- Australia (5):
  - Research Site, East Melbourne
  - Research Site, Kogarah
  - Research Site, Liverpool
  - Research Site, Sydney
  - Research Site, Woolloongabba
- Canada (6):
  - Research Site, Surrey, British Columbia
  - Research Site, Courtice, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Windsor, Ontario
- Germany (10):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Dresden
  - Research Site, Dülmen
  - Research Site, Frankfurt am Main
  - Research Site, Hanover
  - Research Site, München
  - Research Site, Münster
  - Research Site, Stuttgart-Weilimdorf
  - Research Site, Wuppertal
- Japan (4):
  - Research Site, Nakano
  - Research Site, Shibuya-ku
  - Research Site, Shinjuku-ku
  - Research Site, Yokohama
- Poland (5):
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw

REFERENCES:
- [Derived] Silverberg JI, Guttman-Yassky E, Gooderham M, Worm M, Rippon S, O'Quinn S, van der Merwe R, Kragh N, Kurbasic A, Wollenberg A. Health-related quality of life with tralokinumab in moderate-to-severe atopic dermatitis: A phase 2b randomized study. Ann Allergy Asthma Immunol. 2021 May;126(5):576-583.e4. doi: 10.1016/j.anai.2020.12.004. Epub 2020 Dec 15. PMID 33333295
- [Derived] Wollenberg A, Howell MD, Guttman-Yassky E, Silverberg JI, Kell C, Ranade K, Moate R, van der Merwe R. Treatment of atopic dermatitis with tralokinumab, an anti-IL-13 mAb. J Allergy Clin Immunol. 2019 Jan;143(1):135-141. doi: 10.1016/j.jaci.2018.05.029. Epub 2018 Jun 12. PMID 29906525

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 299 participants participated in the study at 55 sites worldwide, including 24 sites in the United States of America, 8 sites in Germany, 6 sites each in Japan, Poland, and Canada, and 5 sites in Australia.
Pre-assignment Details: 95 participants were considered screen failures and 204 participants were randomized and treated in the study.
Groups:
- Placebo: Placebo matched to Tralokinumab was administered subcutaneously to participants once every 2 Weeks (Q2W) for 12 weeks.
- Tralokinumab Dose 1: Tralokinumab Dose 1 was administered subcutaneously to participants once every 2 Weeks (Q2W) for 12 weeks.
- Tralokinumab Dose 2: Tralokinumab Dose 2 was administered subcutaneously to participants once every 2 Weeks (Q2W) for 12 weeks.
- Tralokinumab Dose 3: Tralokinumab Dose 3 was administered subcutaneously to participants once every 2 Weeks (Q2W) for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3
Started | 51 | 50 | 51 | 52
Completed | 39 | 40 | 43 | 48
Not Completed | 12 | 10 | 8 | 4
Not completed — Lost to Follow-up | 2 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 9 | 5 | 5 | 3
Not completed — Other | 1 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized and treated participants, grouped according to assigned treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3 | Total
Number analyzed (Participants) | 51 | 50 | 51 | 52 | 204
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.4 (14.5) | 39.1 (15.1) | 37.1 (14.0) | 35.7 (14.6) | 37.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 21 | 25 | 19 | 94
  Male | 22 | 29 | 26 | 33 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 4 | 11
  Not Hispanic or Latino | 49 | 48 | 48 | 48 | 193
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 10 | 11 | 8 | 16 | 45
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 8 | 4 | 10 | 7 | 29
  White | 31 | 33 | 33 | 28 | 125
  More than one race | 1 | 1 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Week 12
Description: EASI evaluates 4 natural anatomical regions for severity and extent of key disease signs and focuses on the key acute and chronic signs of inflammation (erythema, induration/papulation, excoriation, and lichenification). The maximum total score is 72, with higher values indicating more severe disease. The data presented here is Adjusted mean change after excluding the data from participants who took prohibited medications.
Time Frame: Baseline (Day 1) and Week 12
Population: The intent-to-treat (ITT) population included all randomized and treated participants, grouped according to assigned treatment. Here, the category "Number Analyzed" is number of participants analyzed for this outcome measure.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3
Number analyzed (Participants) | 51 | 50 | 51 | 52
units on a scale | -10.78 (1.398) | -13.67 (1.386) | -15.14 (1.361) | -15.72 (1.334)
Statistical Analysis 1: Comparison: Placebo vs Tralokinumab Dose 1; Test type: Superiority; p = 0.143, Mixed Model Repeated Measures Analysis; Adjusted Mean Difference = -2.89, 95% CI 2-sided [-6.78 to 0.99], Standard Error of Mean 1.968
Statistical Analysis 2: Comparison: Placebo vs Tralokinumab Dose 2; Test type: Superiority; p = 0.027, Mixed Model Repeated Measures Analysis; Adjusted Mean Difference = -4.36, 95% CI 2-sided [-8.22 to -0.51], Standard Error of Mean 1.951
Statistical Analysis 3: Comparison: Placebo vs Tralokinumab Dose 3; Test type: Superiority; p = 0.011, Mixed Model Repeated Measures Analysis; Adjusted Mean Difference = -4.94, 95% CI 2-sided [-8.76 to -1.13], Standard Error of Mean 1.932

2. Primary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) Response of 0 (Clear) or 1 (Almost Clear) and at Least a 2-Grade Reduction From Baseline at Week 12
Description: The IGA allows investigators to assess overall disease severity at one given time point and consists of a 6-point severity scale from clear to very severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease, and 5 = very severe disease). A participant has IGA response if they achieve a score of 0 (clear) or 1 (almost clear) and at least a 2-grade reduction from baseline.
Time Frame: Week 12
Population: The ITT population included all randomized and treated participants, grouped according to assigned treatment. Here, the category "Number Analyzed" is number of participants analyzed for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3
Number analyzed (Participants) | 51 | 50 | 51 | 52
Percentage of participants | 11.8 | 11.6 | 19.5 | 26.7
Statistical Analysis 1: Comparison: Placebo vs Tralokinumab Dose 1; Test type: Superiority; p = 0.974, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.29 to 3.32]
Statistical Analysis 2: Comparison: Placebo vs Tralokinumab Dose 2; Test type: Superiority; p = 0.281, Regression, Logistic; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.61 to 5.65]
Statistical Analysis 3: Comparison: Placebo vs Tralokinumab Dose 3; Test type: Superiority; p = 0.061, Regression, Logistic; Odds Ratio (OR) = 2.83, 95% CI 2-sided [0.95 to 8.37]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) present at baseline that worsened in intensity after administration of investigational product or events absent at baseline that emerged after administration of study drug until Week 22. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening situation (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received Tralokinumab. Treatment-emergent adverse events between administration of investigational product and Week 22 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: From Study Drug Administration (Day 1) to Week 22
Population: As-treated population included all treated participants, grouped according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3
Number analyzed (Participants) | 51 | 50 | 51 | 52
Participants
  TEAEs | 31 | 36 | 35 | 30
  TESAEs | 1 | 3 | 2 | 0

4. Secondary Outcome: Number of Participants With Vital Signs and Physical Examination Abnormalities Reported as Treatment Emergent Adverse Events
Description: Vital sign parameters included blood pressure, temperature, pulse rate, and respiratory rate. TEAEs were present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug until Week 22.
Time Frame: From Study Drug Administration (Day 1) to Week 22
Population: As-treated population included all treated participants, grouped according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3
Number analyzed (Participants) | 51 | 50 | 51 | 52
Participants
  Blood pressure increased | 0 | 1 | 1 | 0
  Pyrexia | 1 | 0 | 1 | 0
  Acute coronary syndrome | 0 | 1 | 0 | 0
  Angina pectoris | 1 | 0 | 0 | 0
  Hypertension | 0 | 0 | 1 | 0
  Pallor | 0 | 0 | 0 | 1

5. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as Treatment Emergent Adverse Events
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as an adverse event. Treatment-emergent adverse events between administration of investigational product and Week 22 that were absent before treatment or that worsened relative to pre-treatment state. Laboratory evaluations (haematology, serum chemistry and urinalysis) of blood and urine samples were performed.
Time Frame: From Study Drug Administration (Day 1) to Week 22
Population: As-treated population included all treated participants, grouped according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3
Number analyzed (Participants) | 51 | 50 | 51 | 52
Participants
  Anaemia | 0 | 1 | 0 | 0
  Lymphopenia | 1 | 0 | 0 | 0
  Alanine aminotransferase increased | 0 | 1 | 0 | 0
  Aspartate aminotransferase increased | 0 | 1 | 0 | 0
  Blood alkaline phosphatase increased | 0 | 0 | 1 | 0
  Blood creatinine increased | 0 | 1 | 0 | 0
  Blood immunoglobulin E increased | 0 | 0 | 1 | 0
  Gamma-glutamyltransferase increased | 0 | 1 | 0 | 0
  Hepatic function abnormal | 0 | 1 | 0 | 0
  Hyperbilirubinaemia | 1 | 0 | 0 | 0
  Liver function test abnormal | 0 | 0 | 1 | 0
  Glycosuria | 0 | 1 | 0 | 0
  Leukocyturia | 1 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities Reported as Treatment Emergent Adverse Events
Description: AEs observed in participants with clinically significant ECG abnormalities were assessed. ECG parameters included heart rate, RR, PR, QRS and QT intervals. Treatment-emergent adverse events between administration of investigational product and Week 22 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: From Study Drug Administration (Day 1) to Week 22
Population: As-treated population included all treated participants, grouped according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3
Number analyzed (Participants) | 51 | 50 | 51 | 52
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Adjusted Percentage of Participants Achieving 50 Percent (%) Reduction From Baseline in Eczema Area and Severity Index (EASI) at Week 12
Description: EASI50 responder is defined as a participant who achieves at least a 50% reduction in EASI score from baseline. Data from participants who took prohibited medications were excluded from this analysis and a last observation carried forward (LOCF) analysis was used.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3
Number analyzed (Participants) | 51 | 50 | 51 | 52
Percentage of participants | 51.9 | 54.3 | 67.3 | 73.4

8. Secondary Outcome: Absolute Change From Baseline in Scoring of Atopic Dermatitis (SCORAD) at Week 12
Description: The SCORAD is a clinical tool for assessing the severity (that is, extent, intensity) of atopic dermatitis (AD). The tool evaluates the extent and intensity of the AD lesions, along with participant symptoms. The maximum total score is 103, with higher values indicating more severe disease. The data presented here is Adjusted mean change after excluding the data from participants who took prohibited medications.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3
Number analyzed (Participants) | 51 | 50 | 51 | 52
units on a scale | -16.67 (2.224) | -21.97 (2.204) | -26.09 (2.168) | -26.50 (2.123)

9. Secondary Outcome: Adjusted Percentage of Participants Achieving 50 Percent (%) Reduction From Baseline in SCORAD at Week 12
Description: SCORAD 50 responder is defined as a participant who achieves at least a 50% reduction in SCORAD score from baseline. Data from participants who took prohibited medications were excluded from this analysis and a LOCF analysis was used.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3
Number analyzed (Participants) | 51 | 50 | 51 | 52
Percentage of participants | 19.5 | 26.9 | 44.2 | 44.1

10. Secondary Outcome: Change From Baseline in Pruritus Numeric Rating Scale (NRS) (7-day Mean Score) at Week 12
Description: Pruritus assessed using an NRS (0 - 10) with 0= no itch and 10= worst imaginable itch. Daily pruritus assessments were summarized as weekly peak score and a change from baseline in weekly peak score was calculated. The data presented here is Adjusted mean change after excluding the data from participants who took prohibited medications.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3
Number analyzed (Participants) | 51 | 50 | 51 | 52
units on a scale | -1.03 (0.270) | -1.80 (0.266) | -1.59 (0.260) | -2.17 (0.256)

ADVERSE EVENTS:
Time Frame: From Study Drug Administration (Day 1) to Week 22
Arm/Group | Placebo | Tralokinumab Dose 1 | Tralokinumab Dose 2 | Tralokinumab Dose 3
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/50 | 0/51 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/51 | 3/50 | 2/51 | 0/52
Other Adverse Events (participants affected / at risk) | 15/51 | 20/50 | 21/51 | 22/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | Tralokinumab Dose 1 (N=50) | Tralokinumab Dose 2 (N=51) | Tralokinumab Dose 3 (N=52)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | Tralokinumab Dose 1 (N=50) | Tralokinumab Dose 2 (N=51) | Tralokinumab Dose 3 (N=52)
Nasopharyngitis (Infections and infestations) | 6 (9) | 11 (12) | 8 (9) | 13 (20)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 5 (7) | 6 (9) | 4 (6)
Headache (Nervous system disorders) | 2 (3) | 3 (6) | 4 (4) | 4 (4)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3) | 3 (4) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.